# Standard Model Consent

Phase II trial of carboplatin and bevacizumab for the treatment of recurrent low-grade and anaplastic supratentorial, infratentorial and spinal cord ependymoma in adults

Subtitle: Phase II Ependymoma

Study 16C0009

Version - Amendment D, May 7, 2019

IRB approval - June 18, 2019

#### Informed Consent

### INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Phase II trial of carboplatin and bevacizumab for the treatment of recurrent low-grade and anaplastic supratentorial, infratentorial and spinal cord ependymoma in adults

Subtitle: Phase II Ependymoma

Study Chair: (insert name of local PI)

Participant's Name

Medical Record Number

You are being asked to take part in this clinical research study at <u>(insert site name)</u>. This consent and authorization form explains why this research study is being done and what your role will be if you choose to take part. This form also describes the possible risks connected with being in this study. After reviewing this information with the person responsible for your enrollment, you should know enough to be able to make an informed decision on whether you want to take part in the study.

You are being asked to take part in this study because you have a brain or spinal cord tumor called an ependymoma that is recurrent (has returned after treatment).

#### PURPOSE OF STUDY

The goal of this clinical research study is to learn if the combination of bevacizumab and carboplatin can help to control recurrent ependymoma. The safety of this drug combination will also be studied.

### **DESCRIPTION OF STUDY**

Study Drugs

**Carboplatin** is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

**Bevacizumab** is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. If some of these tests have been performed within the past 14 days, they may not need to be repeated. The following tests and procedures will be performed:

- Your complete medical history will be recorded, including any drugs you may have taken and/or be taking.
- You will have a complete physical exam, including measurement of your height, weight, and vital signs (heart rate, temperature, breathing rate, and blood pressure).

- You will be asked how well you are able to perform the normal activities of daily living (performance status).
- You will have a neurological exam (tests to check the functioning of your nervous system, including tests of your balance and reflexes). You will also be asked how well you are able to perform tasks like remembering, communicating, and following simple instructions. This should take about 20 minutes to complete.
- Blood (about 2-3 tablespoons) will be drawn for routine tests. This routine blood draw will also include a pregnancy test if you are able to become pregnant. To take part in this study, you must not be pregnant.
- Blood (about 1 teaspoon) will be drawn to check your blood's ability to clot.
- Urine will be collected to check your kidney function.
- You will have a magnetic resonance imaging (MRI) scan or computed tomography (CT) scan of the head and/or spine to check the status of the disease.
- You will complete a questionnaire about your quality of life. The questionnaire should take about 5 minutes to complete.
- Tumor tissue left over from a previous procedure (such as disease diagnosis slides or tumor tissue leftover from a previous biopsy) will be collected to confirm your diagnosis and to test for biomarkers.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

# **Study Drug Administration**

If you are found to be eligible to take part in this study, you will receive carboplatin by vein over 30 minutes on Day 1 of each 28-day cycle. You will receive bevacizumab by vein over 90 minutes on Days 1 and 15 of each cycle.

### **Study Visits**

### Every 2 weeks:

• Blood (about 1 - 2 teaspoons) will be drawn for routine tests

### Every 4 weeks:

- Urine will be collected to check your kidney function.
- You will be asked about any drugs you may be taking and if you have had any side effects.

### Every 8 weeks:

- Your medical history will be recorded.
- You will have a physical exam, including measurement of your vital signs.
- You will have a neurological exam.
- Your performance status will be recorded.
- You will complete the quality of life questionnaire.
- You will have an MRI scan or CT scan of the head and/or spine to check the status of the disease.

At any time during the study, extra tests may be performed if the doctor thinks they are needed for your safety. The study doctor will tell you more about any extra tests.

# **Length of Study**

You will receive up to 6 cycles of the study drug combination. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

If the disease has not gotten worse after 6 cycles of receiving the study drug combination, you will be able to continue receiving bevacizumab alone for as long as the doctor thinks it is in your best interest. You will continue to follow the same study visit schedule detailed above.

## Long-Term Follow-up

If you go off study because the disease got worse or you experienced intolerable side effects, the study staff will call you every 3 months from then on to check your health. Each phone call should take about 5 minutes.

This is an investigational study. Carboplatin is FDA approved and commercially available for the treatment of advanced ovarian cancer. Bevacizumab is FDA approved and commercially available for the treatment of glioblastoma (a type of brain tumor). The use of these drugs in combination in ependymoma is investigational.

You and/or your insurance provider will be responsible for the costs of carboplatin and bevacizumab.

Up to 46 patients will take part in this study. Up to (insert local accrual ceiling) will be enrolled at (insert site name).

## RISKS, SIDE EFFECTS, AND DISCOMFORTS TO PARTICIPANTS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases, side effects may be serious, long-lasting or permanent, and may even cause death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs.

Carboplatin and bevacizumab may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# **Carboplatin Side Effects**

| abnormal salts, minerals,<br>and/or acids in the blood | 1 - 1 1 1 4 - ( 1 | abnormal liver tests (possible liver damage) |
|---|---|---|
|---|---|---|

#### Informed Consent

### INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Phase II trial of carboplatin and bevacizumab for the treatment of recurrent low-grade and anaplastic supratentorial, infratentorial and spinal cord ependymoma in adults

Subtitle: Phase II Ependymoma

Study Chair: (insert name of local PI)

Participant's Name

Medical Record Number

You are being asked to take part in this clinical research study at <u>(insert site name)</u>. This consent and authorization form explains why this research study is being done and what your role will be if you choose to take part. This form also describes the possible risks connected with being in this study. After reviewing this information with the person responsible for your enrollment, you should know enough to be able to make an informed decision on whether you want to take part in the study.

You are being asked to take part in this study because you have a brain or spinal cord tumor called an ependymoma that is recurrent (has returned after treatment).

#### PURPOSE OF STUDY

The goal of this clinical research study is to learn if the combination of bevacizumab and carboplatin can help to control recurrent ependymoma. The safety of this drug combination will also be studied.

### **DESCRIPTION OF STUDY**

Study Drugs

**Carboplatin** is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

**Bevacizumab** is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. If some of these tests have been performed within the past 14 days, they may not need to be repeated. The following tests and procedures will be performed:

- Your complete medical history will be recorded, including any drugs you may have taken and/or be taking.
- You will have a complete physical exam, including measurement of your height, weight, and vital signs (heart rate, temperature, breathing rate, and blood pressure).

- You will be asked how well you are able to perform the normal activities of daily living (performance status).
- You will have a neurological exam (tests to check the functioning of your nervous system, including tests of your balance and reflexes). You will also be asked how well you are able to perform tasks like remembering, communicating, and following simple instructions. This should take about 20 minutes to complete.
- Blood (about 2-3 tablespoons) will be drawn for routine tests. This routine blood draw will also include a pregnancy test if you are able to become pregnant. To take part in this study, you must not be pregnant.
- Blood (about 1 teaspoon) will be drawn to check your blood's ability to clot.
- Urine will be collected to check your kidney function.
- You will have a magnetic resonance imaging (MRI) scan or computed tomography (CT) scan of the head and/or spine to check the status of the disease.
- You will complete a questionnaire about your quality of life. The questionnaire should take about 5 minutes to complete.
- Tumor tissue left over from a previous procedure (such as disease diagnosis slides or tumor tissue leftover from a previous biopsy) will be collected to confirm your diagnosis and to test for biomarkers.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

# **Study Drug Administration**

If you are found to be eligible to take part in this study, you will receive carboplatin by vein over 30 minutes on Day 1 of each 28-day cycle. You will receive bevacizumab by vein over 90 minutes on Days 1 and 15 of each cycle.

### **Study Visits**

### Every 2 weeks:

• Blood (about 1 - 2 teaspoons) will be drawn for routine tests

### Every 4 weeks:

- Urine will be collected to check your kidney function.
- You will be asked about any drugs you may be taking and if you have had any side effects.

### Every 8 weeks:

- Your medical history will be recorded.
- You will have a physical exam, including measurement of your vital signs.
- You will have a neurological exam.
- Your performance status will be recorded.
- You will complete the quality of life questionnaire.
- You will have an MRI scan or CT scan of the head and/or spine to check the status of the disease.

At any time during the study, extra tests may be performed if the doctor thinks they are needed for your safety. The study doctor will tell you more about any extra tests.

# **Length of Study**

You will receive up to 6 cycles of the study drug combination. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

If the disease has not gotten worse after 6 cycles of receiving the study drug combination, you will be able to continue receiving bevacizumab alone for as long as the doctor thinks it is in your best interest. You will continue to follow the same study visit schedule detailed above.

## Long-Term Follow-up

If you go off study because the disease got worse or you experienced intolerable side effects, the study staff will call you every 3 months from then on to check your health. Each phone call should take about 5 minutes.

This is an investigational study. Carboplatin is FDA approved and commercially available for the treatment of advanced ovarian cancer. Bevacizumab is FDA approved and commercially available for the treatment of glioblastoma (a type of brain tumor). The use of these drugs in combination in ependymoma is investigational.

You and/or your insurance provider will be responsible for the costs of carboplatin and bevacizumab.

Up to 46 patients will take part in this study. Up to (insert local accrual ceiling) will be enrolled at (insert site name).

## RISKS, SIDE EFFECTS, AND DISCOMFORTS TO PARTICIPANTS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases, side effects may be serious, long-lasting or permanent, and may even cause death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs.

Carboplatin and bevacizumab may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# **Carboplatin Side Effects**

| abnormal salts, minerals,<br>and/or acids in the blood | 1 - 1 1 1 4 - ( 1 | abnormal liver tests (possible liver damage) |
|---|---|---|
|---|---|---|

#### Informed Consent

### INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Phase II trial of carboplatin and bevacizumab for the treatment of recurrent low-grade and anaplastic supratentorial, infratentorial and spinal cord ependymoma in adults

Subtitle: Phase II Ependymoma

Study Chair: (insert name of local PI)

Participant's Name

Medical Record Number

You are being asked to take part in this clinical research study at <u>(insert site name)</u>. This consent and authorization form explains why this research study is being done and what your role will be if you choose to take part. This form also describes the possible risks connected with being in this study. After reviewing this information with the person responsible for your enrollment, you should know enough to be able to make an informed decision on whether you want to take part in the study.

You are being asked to take part in this study because you have a brain or spinal cord tumor called an ependymoma that is recurrent (has returned after treatment).

#### PURPOSE OF STUDY

The goal of this clinical research study is to learn if the combination of bevacizumab and carboplatin can help to control recurrent ependymoma. The safety of this drug combination will also be studied.

### **DESCRIPTION OF STUDY**

Study Drugs

**Carboplatin** is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

**Bevacizumab** is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. If some of these tests have been performed within the past 14 days, they may not need to be repeated. The following tests and procedures will be performed:

- Your complete medical history will be recorded, including any drugs you may have taken and/or be taking.
- You will have a complete physical exam, including measurement of your height, weight, and vital signs (heart rate, temperature, breathing rate, and blood pressure).

# **Length of Study**

You will receive up to 6 cycles of the study drug combination. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

If the disease has not gotten worse after 6 cycles of receiving the study drug combination, you will be able to continue receiving bevacizumab alone for as long as the doctor thinks it is in your best interest. You will continue to follow the same study visit schedule detailed above.

## Long-Term Follow-up

If you go off study because the disease got worse or you experienced intolerable side effects, the study staff will call you every 3 months from then on to check your health. Each phone call should take about 5 minutes.

This is an investigational study. Carboplatin is FDA approved and commercially available for the treatment of advanced ovarian cancer. Bevacizumab is FDA approved and commercially available for the treatment of glioblastoma (a type of brain tumor). The use of these drugs in combination in ependymoma is investigational.

You and/or your insurance provider will be responsible for the costs of carboplatin and bevacizumab.

Up to 46 patients will take part in this study. Up to (insert local accrual ceiling) will be enrolled at (insert site name).

## RISKS, SIDE EFFECTS, AND DISCOMFORTS TO PARTICIPANTS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases, side effects may be serious, long-lasting or permanent, and may even cause death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs.

Carboplatin and bevacizumab may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# **Carboplatin Side Effects**

| abnormal salts, minerals,<br>and/or acids in the blood | 1 - 1 1 1 4 - ( 1 | abnormal liver tests (possible liver damage) |
|---|---|---|
|---|---|---|

| (possible weakness, | • pain | abnormal kidney test |
|------------------------------|--------|-------------------------|
| swelling, fatigue, low blood | | (possible kidney damage |
| pressure, organ failure, | | |
| heart problems, changes in | | |
| mental status, and/or | | |
| seizure) | | |

| • | nerve damage (possible | ' |
|---|-----------------------------|---|
| | numbness, pain, and/or loss | ' |
| | of motor function) | • |
| | 1 1 1 / 1 1 1 | |

- hair loss (partial or total)
- abdominal pain
- nausea

- constipation
- diarrhea
- abnormal taste
- mouth blisters/sores (possible difficulty swallowing)
- weakness
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- allergic reaction
- infection

## Rare but serious (occurring in fewer than 3% of patients)

- high blood pressure
- low blood pressure (possible dizziness/fainting)
- heart failure
- stroke
- dehydration
- blood vessel blockage
- anemia due to destruction of red blood cells
- multiple blood clots (possible organ dysfunction and/or failure)
- reduced blood supply to the arms and legs
- visual problems
- blindness
- hearing loss

- difficulty breathing due to narrowing of the airways
- tissue death at the injection site caused by drug leakage
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

Carboplatin may rarely cause you to develop another type of cancer.

### **Bevacizumab Side Effects**

- high blood pressure
- blood clots in a vein (possible pain, swelling, and/or redness)
- pain
- nerve damage (loss of sensory function)
- headache
- dizziness
- fatigue
- hair loss (partial or total)
- abdominal pain

- loss of appetite
- constipation
- diarrhea
- mouth blisters/sores (possible difficulty swallowing)
- digestive system bleeding
- upset stomach
- vomiting
- abnormal taste

- failure of the ovaries to produce hormones, which may be permanent (possible stopped menstrual cycle)
- bleeding
- nosebleed
- low white blood cell counts
- difficulty breathing
- weakness

| abnormal kidney test (possible kidney) |
|--------------------------------------------|
| damage) |

- blood clots in an artery (possible organ damage such as stroke and/or heart attack)
- low blood pressure (possible dizziness/fainting)
- heart failure
- fainting
- bleeding in the brain and/or spinal cord
- stroke
- difficulty walking
- dry skin
- skin sores
- opening of a wound

- shedding and scaling of the skin (possible fatal loss of bodily fluids)
- change of skin color
- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)
- dehydration
- gas
- dry mouth
- hole in the intestines (possibly leaking contents into the abdomen)
- bleeding gums

- inflammation or paralysis of the intestines
- weight loss
- nausea
- uterine and/or vaginal bleeding
- low platelet cell counts
- pain (back/muscle)
- voice changes
- runny nose
- lung inflammation (possible difficulty breathing)
- infusion reaction (possible chills and/or hives)

# Rare but serious (occurring in fewer than 3% of patients)

- severe heart problems
- heart attack
- chest pain due to heart trouble
- severe increase in blood pressure (possible stroke)
- brain injury that may be reversible (possible headache, confusion, seizures, and/or vision loss)
- decreased brain function due to high blood pressure
- decreased blood flow to part of the bowel (possibly causing death of tissue)
- bleeding around the brain
- temporary stroke symptoms
- intestinal blockage

- stomach and/or small intestine ulcer
- vein blockage in the abdomen
- hole in the gall bladder (possible abdominal pain, gall stones, nausea, and/or infection)
- hole in the bladder
- destruction of red blood cells
- low red blood cell counts
- bone destruction
   (including destruction of
   the jaw bone)
- inflammation inside the eye
- blurry vision

- deafness
- kidney failure
- decreased kidney function (possible kidney failure)
- coughing up blood
- increased blood pressure in the lungs (possible difficulty breathing and/or heart failure)
- blockage in the lung (possible pain, shortness of breath, and/or failure to breathe)
- abnormal hole inside the nose
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

| <ul> <li>increased pressure in the eye (possible pain and/or blurry vision)</li> <li>detached retina (possible</li> </ul> |
|---|
| partial blindness) |

Bevacizumab may rarely cause an abnormal opening that develops between one area of the body and another (for example, an abnormal connection and opening in one or more places between the trachea [breathing tube] and esophagus, which may interfere with swallowing, digestion, and/or choking). This may result in death.

Rarely (in about 1-2% of patients), bevacizumab may cause bleeding in the brain in patients who have received bevacizumab for the treatment of primary brain tumors. You will be monitored for this complication and removed from the study if this were to occur.

If you are taking Coumadin (warfarin) or other blood-thinning drugs, you may be at higher risk of blood clots and/or bleeding.

Using **the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns after completing the questionnaire, you are encouraged to contact your doctor or the study chair.

This study may involve unpredictable risks to the participants.

### **Pregnancy Related Risks**

Because taking part in this study can result in risks to an unborn or breastfeeding baby, you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you are able to become pregnant or father a child, you must use acceptable birth control while on study and for 1 month after the last dose of study drug(s). Medically acceptable birth control types include approved hormonal birth control (such as birth control pills, Depo-Provera, or Lupron Depot), barrier methods (such as a condom or diaphragm) with spermicide, or intrauterine device (IUD). Talk to the study doctor about acceptable methods of birth control.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant may result in your removal from this study.

| (possible weakness, | • pain | abnormal kidney test |
|------------------------------|--------|-------------------------|
| swelling, fatigue, low blood | | (possible kidney damage |
| pressure, organ failure, | | |
| heart problems, changes in | | |
| mental status, and/or | | |
| seizure) | | |

| • | nerve damage (possible | • | con |
|---|------------------------------|---|-----|
| | numbness, pain, and/or loss | • | dia |
| | of motor function) | • | abn |
| • | hair loss (partial or total) | • | mo |

- abdominal pain
- nausea

- nstipation
- arrhea
- normal taste
- outh blisters/sores (possible difficulty swallowing)
- weakness
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- allergic reaction
- infection

## Rare but serious (occurring in fewer than 3% of patients)

- high blood pressure
- low blood pressure (possible dizziness/fainting)
- heart failure
- stroke
- dehydration
- blood vessel blockage
- anemia due to destruction of red blood cells
- multiple blood clots (possible organ dysfunction and/or failure)
- reduced blood supply to the arms and legs
- visual problems
- blindness
- hearing loss

- difficulty breathing due to narrowing of the airways
- tissue death at the injection site caused by drug leakage
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

Carboplatin may rarely cause you to develop another type of cancer.

### **Bevacizumab Side Effects**

- high blood pressure
- blood clots in a vein (possible pain, swelling, and/or redness)
- nerve damage (loss of sensory function)
- headache
- dizziness
- fatigue
- hair loss (partial or total)
- abdominal pain

- loss of appetite
- constipation
- diarrhea
- mouth blisters/sores (possible difficulty swallowing)
- digestive system bleeding
- upset stomach
- vomiting
- abnormal taste

- failure of the ovaries to produce hormones, which may be permanent (possible stopped menstrual cycle)
- bleeding
- nosebleed
- low white blood cell counts
- difficulty breathing
- weakness

| abnormal kidney test (possible kidney) |
|--------------------------------------------|
| damage) |

- blood clots in an artery (possible organ damage such as stroke and/or heart attack)
- low blood pressure (possible dizziness/fainting)
- heart failure
- fainting
- bleeding in the brain and/or spinal cord
- stroke
- difficulty walking
- dry skin
- skin sores
- opening of a wound

- shedding and scaling of the skin (possible fatal loss of bodily fluids)
- change of skin color
- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)
- dehydration
- gas
- dry mouth
- hole in the intestines (possibly leaking contents into the abdomen)
- bleeding gums

- inflammation or paralysis of the intestines
- weight loss
- nausea
- uterine and/or vaginal bleeding
- low platelet cell counts
- pain (back/muscle)
- voice changes
- runny nose
- lung inflammation (possible difficulty breathing)
- infusion reaction (possible chills and/or hives)

# Rare but serious (occurring in fewer than 3% of patients)

- severe heart problems
- heart attack
- chest pain due to heart trouble
- severe increase in blood pressure (possible stroke)
- brain injury that may be reversible (possible headache, confusion, seizures, and/or vision loss)
- decreased brain function due to high blood pressure
- decreased blood flow to part of the bowel (possibly causing death of tissue)
- bleeding around the brain
- temporary stroke symptoms
- intestinal blockage

- stomach and/or small intestine ulcer
- vein blockage in the abdomen
- hole in the gall bladder (possible abdominal pain, gall stones, nausea, and/or infection)
- hole in the bladder
- destruction of red blood cells
- low red blood cell counts
- bone destruction
   (including destruction of
   the jaw bone)
- inflammation inside the eye
- blurry vision

- deafness
- kidney failure
- decreased kidney function (possible kidney failure)
- coughing up blood
- increased blood pressure in the lungs (possible difficulty breathing and/or heart failure)
- blockage in the lung (possible pain, shortness of breath, and/or failure to breathe)
- abnormal hole inside the nose
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

#### Informed Consent

## INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Phase II trial of carboplatin and bevacizumab for the treatment of recurrent low-grade and anaplastic supratentorial, infratentorial and spinal cord ependymoma in adults

Subtitle: Phase II Ependymoma

Study Chair: (insert name of local PI)

Participant's Name

Medical Record Number

You are being asked to take part in this clinical research study at <u>(insert site name)</u>. This consent and authorization form explains why this research study is being done and what your role will be if you choose to take part. This form also describes the possible risks connected with being in this study. After reviewing this information with the person responsible for your enrollment, you should know enough to be able to make an informed decision on whether you want to take part in the study.

You are being asked to take part in this study because you have a brain or spinal cord tumor called an ependymoma that is recurrent (has returned after treatment).

#### PURPOSE OF STUDY

The goal of this clinical research study is to learn if the combination of bevacizumab and carboplatin can help to control recurrent ependymoma. The safety of this drug combination will also be studied.

### **DESCRIPTION OF STUDY**

Study Drugs

**Carboplatin** is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

**Bevacizumab** is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. If some of these tests have been performed within the past 14 days, they may not need to be repeated. The following tests and procedures will be performed:

- Your complete medical history will be recorded, including any drugs you may have taken and/or be taking.
- You will have a complete physical exam, including measurement of your height, weight, and vital signs (heart rate, temperature, breathing rate, and blood pressure).

- You will be asked how well you are able to perform the normal activities of daily living (performance status).
- You will have a neurological exam (tests to check the functioning of your nervous system, including tests of your balance and reflexes). You will also be asked how well you are able to perform tasks like remembering, communicating, and following simple instructions. This should take about 20 minutes to complete.
- Blood (about 2-3 tablespoons) will be drawn for routine tests. This routine blood draw will also include a pregnancy test if you are able to become pregnant. To take part in this study, you must not be pregnant.
- Blood (about 1 teaspoon) will be drawn to check your blood's ability to clot.
- Urine will be collected to check your kidney function.
- You will have a magnetic resonance imaging (MRI) scan or computed tomography (CT) scan of the head and/or spine to check the status of the disease.
- You will complete a questionnaire about your quality of life. The questionnaire should take about 5 minutes to complete.
- Tumor tissue left over from a previous procedure (such as disease diagnosis slides or tumor tissue leftover from a previous biopsy) will be collected to confirm your diagnosis and to test for biomarkers.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

# **Study Drug Administration**

If you are found to be eligible to take part in this study, you will receive carboplatin by vein over 30 minutes on Day 1 of each 28-day cycle. You will receive bevacizumab by vein over 90 minutes on Days 1 and 15 of each cycle.

### **Study Visits**

### Every 2 weeks:

• Blood (about 1 - 2 teaspoons) will be drawn for routine tests

### Every 4 weeks:

- Urine will be collected to check your kidney function.
- You will be asked about any drugs you may be taking and if you have had any side effects.

### Every 8 weeks:

- Your medical history will be recorded.
- You will have a physical exam, including measurement of your vital signs.
- You will have a neurological exam.
- Your performance status will be recorded.
- You will complete the quality of life questionnaire.
- You will have an MRI scan or CT scan of the head and/or spine to check the status of the disease.

At any time during the study, extra tests may be performed if the doctor thinks they are needed for your safety. The study doctor will tell you more about any extra tests.

# **Length of Study**

You will receive up to 6 cycles of the study drug combination. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

If the disease has not gotten worse after 6 cycles of receiving the study drug combination, you will be able to continue receiving bevacizumab alone for as long as the doctor thinks it is in your best interest. You will continue to follow the same study visit schedule detailed above.

## Long-Term Follow-up

If you go off study because the disease got worse or you experienced intolerable side effects, the study staff will call you every 3 months from then on to check your health. Each phone call should take about 5 minutes.

This is an investigational study. Carboplatin is FDA approved and commercially available for the treatment of advanced ovarian cancer. Bevacizumab is FDA approved and commercially available for the treatment of glioblastoma (a type of brain tumor). The use of these drugs in combination in ependymoma is investigational.

You and/or your insurance provider will be responsible for the costs of carboplatin and bevacizumab.

Up to 46 patients will take part in this study. Up to (insert local accrual ceiling) will be enrolled at (insert site name).

## RISKS, SIDE EFFECTS, AND DISCOMFORTS TO PARTICIPANTS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases, side effects may be serious, long-lasting or permanent, and may even cause death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs.

Carboplatin and bevacizumab may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# **Carboplatin Side Effects**

| abnormal salts, minerals,<br>and/or acids in the blood | 1 - 1 1 1 4 - ( 1 | abnormal liver tests (possible liver damage) |
|---|---|---|
|---|---|---|

| (possible weakness, | • pain | abnormal kidney test |
|------------------------------|--------|-------------------------|
| swelling, fatigue, low blood | | (possible kidney damage |
| pressure, organ failure, | | |
| heart problems, changes in | | |
| mental status, and/or | | |
| seizure) | | |

| • | nerve damage (possible | • | con |
|---|------------------------------|---|-----|
| | numbness, pain, and/or loss | • | dia |
| | of motor function) | • | abn |
| • | hair loss (partial or total) | • | mo |

- abdominal pain
- nausea

- nstipation
- arrhea
- normal taste
- outh blisters/sores (possible difficulty swallowing)
- weakness
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- allergic reaction
- infection

## Rare but serious (occurring in fewer than 3% of patients)

- high blood pressure
- low blood pressure (possible dizziness/fainting)
- heart failure
- stroke
- dehydration
- blood vessel blockage
- anemia due to destruction of red blood cells
- multiple blood clots (possible organ dysfunction and/or failure)
- reduced blood supply to the arms and legs
- visual problems
- blindness
- hearing loss

- difficulty breathing due to narrowing of the airways
- tissue death at the injection site caused by drug leakage
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

Carboplatin may rarely cause you to develop another type of cancer.

### **Bevacizumab Side Effects**

- high blood pressure
- blood clots in a vein (possible pain, swelling, and/or redness)
- nerve damage (loss of sensory function)
- headache
- dizziness
- fatigue
- hair loss (partial or total)
- abdominal pain

- loss of appetite
- constipation
- diarrhea
- mouth blisters/sores (possible difficulty swallowing)
- digestive system bleeding
- upset stomach
- vomiting
- abnormal taste

- failure of the ovaries to produce hormones, which may be permanent (possible stopped menstrual cycle)
- bleeding
- nosebleed
- low white blood cell counts
- difficulty breathing
- weakness

| abnormal kidney test (possible kidney) |
|--------------------------------------------|
| damage) |

- blood clots in an artery (possible organ damage such as stroke and/or heart attack)
- low blood pressure (possible dizziness/fainting)
- heart failure
- fainting
- bleeding in the brain and/or spinal cord
- stroke
- difficulty walking
- dry skin
- skin sores
- opening of a wound

- shedding and scaling of the skin (possible fatal loss of bodily fluids)
- change of skin color
- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)
- dehydration
- gas
- dry mouth
- hole in the intestines (possibly leaking contents into the abdomen)
- bleeding gums

- inflammation or paralysis of the intestines
- weight loss
- nausea
- uterine and/or vaginal bleeding
- low platelet cell counts
- pain (back/muscle)
- voice changes
- runny nose
- lung inflammation (possible difficulty breathing)
- infusion reaction (possible chills and/or hives)

# Rare but serious (occurring in fewer than 3% of patients)

- severe heart problems
- heart attack
- chest pain due to heart trouble
- severe increase in blood pressure (possible stroke)
- brain injury that may be reversible (possible headache, confusion, seizures, and/or vision loss)
- decreased brain function due to high blood pressure
- decreased blood flow to part of the bowel (possibly causing death of tissue)
- bleeding around the brain
- temporary stroke symptoms
- intestinal blockage

- stomach and/or small intestine ulcer
- vein blockage in the abdomen
- hole in the gall bladder (possible abdominal pain, gall stones, nausea, and/or infection)
- hole in the bladder
- destruction of red blood cells
- low red blood cell counts
- bone destruction
   (including destruction of
   the jaw bone)
- inflammation inside the eye
- blurry vision

- deafness
- kidney failure
- decreased kidney function (possible kidney failure)
- coughing up blood
- increased blood pressure in the lungs (possible difficulty breathing and/or heart failure)
- blockage in the lung (possible pain, shortness of breath, and/or failure to breathe)
- abnormal hole inside the nose
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

| <ul> <li>increased pressure in the eye (possible pain and/or blurry vision)</li> <li>detached retina (possible</li> </ul> |
|---|
| partial blindness) |

Bevacizumab may rarely cause an abnormal opening that develops between one area of the body and another (for example, an abnormal connection and opening in one or more places between the trachea [breathing tube] and esophagus, which may interfere with swallowing, digestion, and/or choking). This may result in death.

Rarely (in about 1-2% of patients), bevacizumab may cause bleeding in the brain in patients who have received bevacizumab for the treatment of primary brain tumors. You will be monitored for this complication and removed from the study if this were to occur.

If you are taking Coumadin (warfarin) or other blood-thinning drugs, you may be at higher risk of blood clots and/or bleeding.

Using **the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns after completing the questionnaire, you are encouraged to contact your doctor or the study chair.

This study may involve unpredictable risks to the participants.

### **Pregnancy Related Risks**

Because taking part in this study can result in risks to an unborn or breastfeeding baby, you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you are able to become pregnant or father a child, you must use acceptable birth control while on study and for 1 month after the last dose of study drug(s). Medically acceptable birth control types include approved hormonal birth control (such as birth control pills, Depo-Provera, or Lupron Depot), barrier methods (such as a condom or diaphragm) with spermicide, or intrauterine device (IUD). Talk to the study doctor about acceptable methods of birth control.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant may result in your removal from this study.

| <ul> <li>increased pressure in the eye (possible pain and/or blurry vision)</li> <li>detached retina (possible</li> </ul> |
|---|
| partial blindness) |

Bevacizumab may rarely cause an abnormal opening that develops between one area of the body and another (for example, an abnormal connection and opening in one or more places between the trachea [breathing tube] and esophagus, which may interfere with swallowing, digestion, and/or choking). This may result in death.

Rarely (in about 1-2% of patients), bevacizumab may cause bleeding in the brain in patients who have received bevacizumab for the treatment of primary brain tumors. You will be monitored for this complication and removed from the study if this were to occur.

If you are taking Coumadin (warfarin) or other blood-thinning drugs, you may be at higher risk of blood clots and/or bleeding.

Using **the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns after completing the questionnaire, you are encouraged to contact your doctor or the study chair.

This study may involve unpredictable risks to the participants.

### **Pregnancy Related Risks**

Because taking part in this study can result in risks to an unborn or breastfeeding baby, you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you are able to become pregnant or father a child, you must use acceptable birth control while on study and for 1 month after the last dose of study drug(s). Medically acceptable birth control types include approved hormonal birth control (such as birth control pills, Depo-Provera, or Lupron Depot), barrier methods (such as a condom or diaphragm) with spermicide, or intrauterine device (IUD). Talk to the study doctor about acceptable methods of birth control.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant may result in your removal from this study.

#### POTENTIAL BENEFITS

The study drugs may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

## ALTERNATIVE PROCEDURES OR TREATMENTS

You may choose not to take part in this study. You may choose to receive other treatments for recurrent ependymoma (such as chemotherapy [such as temozolomide], radiation therapy, or a combination of both). You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

### ADDITIONAL INFORMATION

You may ask the study chair any questions you have about this study. You may contact the study chair, *insert local PI name*, at *insert local PI contact information*. You may also contact the Chair of *insert local IRB name* (IRB - a committee that reviews research studies) at *insert local IRB contact information* with any questions that have to do with this study or your rights as a study participant.

Your participation in this research study is strictly voluntary. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor.

This study or your participation in it may be changed or stopped at any time by the study chair, the National Cancer Institute, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP - a regulatory agency that oversees research in humans), or the IRB of *insert local IRB name*.

You will be informed of any new findings that might affect your willingness to continue taking part in the study.

This study is coordinated by The National Cancer Institute, Center for Cancer Research.

### STUDY COSTS AND COMPENSATION

## (Tailor per local institution policy)

If you suffer injury as a direct result of taking part in this study, *insert site name* health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by *insert site name* or the National Cancer Institute for this injury. You may also contact the Chair *insert local IRB name and contact information* with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs, including hospitalization, nausea, vomiting, low blood cell counts, and dehydration. Standard medical care that you receive under this research

study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

### WILL YOUR MEDICAL INFORMATION BE KEPT PRIVATE?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- Insert local IRB name
- National Institute of Health Institutional Review Board

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to the NIH IRB or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases can**not** be recalled and destroyed.

### **CERTIFICATE OF CONFIDENTIALITY**

To help us protect your privacy, we have obtained a Certificate of Confidentiality. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

You should also know that there are several circumstances in which the Certificate does not provide coverage. These include when information:

- will be used for auditing or program evaluation internally by the NIH; or
- must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA).
- is necessary for your medical treatment and you have consented to this disclosure;
- is for other research.

In addition, identifiable, sensitive information protected by this Certificate cannot be admissible as evidence or used for any purpose in any action, suit, or proceeding without your consent.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

### USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

### Notes to consent form authors:

The NCI has recommended that HIPAA regulations be addressed by the local institution. Language pertaining to HIPAA compliance may or may not be included in the local consent form, depending on local institutional policy.

### CONSENT/AUTHORIZATION

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

SIGNATURE OF PARTICIPANT DATE

### PERSON OBTAINING CONSENT

I have discussed this clinical research study with the participant, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation.

SIGNATURE OF STUDY CHAIR OR PERSON AUTHORIZED TO DATE OBTAIN CONSENT